CLINICAL TRIAL: NCT01726933
Title: A Multi-center, Randomized, Double-blind, Three-arm, 16 Week, Adaptive Phase III Clinical Study to Investigate the Efficacy and Safety of LAS41008 vs LASW1835 and vs Placebo in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: LAS41008 in Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Almirall Hermal GmbH (Industry); Harrison Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M41008-1102; 2012-000055-13 (EudraCT Number)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Plaque Psoriasis
Keywords: psoriasis, systemic treatment
MeSH Terms: conditions — Psoriasis | interventions — calcium D-pantothenate, L-cysteine drug combination; Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LAS41008 (Experimental): up to 6 tablets/ day for 16 weeks double blind treatment period, randomized gastric resistant tablet
  Interventions: Drug: LAS41008
- Placebo (Placebo Comparator): up to 6 tablets/ day for 16 weeks randomized, double blind gastric resistant tablet
  Interventions: Drug: Placebo
- LASW1835 (Active Comparator): double blind, randomized gastric resistant tablet up to 6 tablets/ day for 16 weeks
  Interventions: Drug: LASW1835

INTERVENTIONS:
Drug: LAS41008 — gastric resistant tablet, weekly up-titration up to maximal tolerated dosage
  Other Names: Verum
  Arms: LAS41008
Drug: LASW1835 — gastric resistant tablet, weekly up-titration up to maximal tolerated dosage
  Other Names: Fumaderm initial/ Fumaderm
  Arms: LASW1835
Drug: Placebo — gastric resistant tablet, weekly up-titration up to maximal tolerated dosage
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of LAS41008 in comparison to active control and placebo in patients with moderate to severe chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Signed and personally dated written informed consent
2. Male / female
3. Aged 18 years or older
4. With a diagnosis of chronic plaque psoriasis for at least 12 months before enrollment in the study
5. With the severity of psoriasis defined as moderate to severe, as reflected in meeting all the following criteria:

   * PASI > 10
   * BSA (body surface area) > 10 %
   * PGA moderate to severe
6. With general good health, or a stable medical condition not considered likely to interfere with the conduct of the clinical study, as determined by the investigator based upon results of medical history, laboratory results and physical examination
7. Prior therapy with systemic drugs for psoriasis or naïve to systemic treatment but identified as a candidate for systemic treatment.
8. With a complete record of at least 12 months of other previous topical and systemic treatments, if any
9. Adhering to the following wash-out periods Topical treatment Wash-out Period Corticosteroids Vitamin A analogues Vitamin D analogues Anthracene derivatives Tar Salicylic acid preparations 2 weeks Systemic treatment Biologics with antipsoriatic activity 3 months Conventional systemic antipsoriatic drugs and phototherapy 1 month Immunosuppressive medication (if not covered by any of the above treatments) Cytostatics 6 months Medications with known harmful influences on the kidneys 5 x halftime
10. For females of child-bearing potential: a negative serum pregnancy test at screening and willing to use highly effective methods of birth control during the study period and for 60 days after the last dose of investigational product. Additionally they must agree to have pregnancy tests while on study medication. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomized partner. Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years.
11. Males (including those who have had vasectomy) must agree to use barrier contraception while on study medication
12. Willing to keep sun exposure reasonably constant and not to use tanning booths or other UV light sources for the duration of the trial

Exclusion Criteria:

1. For females: pregnant or lactating
2. With a diagnosis of guttate, erythrodermic or pustular psoriasis
3. With a hematological abnormality as follows: platelet count < 100,000/mm3, WBC count < 3,000 cells/ mm3, lymphocyte count < 1.000/µl, hemoglobin, hematocrit, or red blood cell count outside 30 % of the upper or lower limits of normal for the lab
4. With a history of malignancies except for non melanoma skin cancer
5. Suffering from significant gastrointestinal problems (ulcers, diarrhea, etc.)
6. Known to have significant renal impairment
7. Are detected to have abnormal liver enzymes >2x the upper limit of the normal range
8. With active infectious disease
9. On systemic therapy with drugs that may interfere with the investigational products taken within the defined wash-out period
10. With a history of alcohol or drug abuse
11. Known HIV-positive status or suffering from any other immunosuppressive disease
12. Known to be hypersensitive to ingredients of the investigational products
13. Previous enrolled in this study or participating in any other drug investigational trial within the 30 days (or five half-lives whichever is longer) prior to enrolment.
14. Not willing to give consent for transmission of personal "pseudonymised" data
15. Unable to comply with the requirements of the study or who in the opinion of the investigator should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
PASI 75 | 16 weeks
  Reduction of PASI by 75% from baseline to week 16
Physician Global Assessment, PGA | 16 weeks
  Change in PGA from baseline to week 16

SECONDARY OUTCOMES:
Body Surface Area, BSA | 16 weeks
  Change in BSA from baseline to week 3, 8, 16 and follow up
Dermatological Life Quality Index, DLQI | 16 weeks
  Change in DLQI from baseline to week 3, 8, 16 and follow up
PASI 75 | week 3 and 8
  Change in PASI 75 from baseline to week 3 and 8 and follow up
PGA | week 3 and 8
  Change in PGA from baseline to week 3 and 8 and follow up
Adverse events | ongoing
  Ongoing safety profile over the course of the study (treatment phase and follow up)

OTHER OUTCOMES:
Patient Benefit Index, PBI | week 16
  Calculation of individual benefit from therapy, assessed by patient at week 16 and in follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Mrowietz, MD, Prof, Principal Investigator — University Medical Center, Schleswig-Holstein, Department of Dermatology, Schittenhelmstr. 7, 24105 Kiel, Germany
Locations (4):
- Investigatives site names will not be disclosed to avoid competitive information. Specify at least one site as follows: Almirall Investigative Site, Various, Austria
- Investigatives site names will not be disclosed to avoid competitive information. Specify at least one site as follows: Almirall Investigative Site, Various, Germany
- Investigatives site names will not be disclosed to avoid competitive information. Specify at least one site as follows: Almirall Investigative Site, Various, Netherlands
- Investigatives site names will not be disclosed to avoid competitive information. Specify at least one site as follows:Almirall Investigative Site #, Various, Poland

REFERENCES:
- [Derived] Warren RB, Barker JNW, Van de Kerkhof P, Reich K, Mrowietz U. Switching from a fumaric acid ester mixture to dimethylfumarate monotherapy in psoriasis. J Eur Acad Dermatol Venereol. 2019 Oct;33(10):e352-e353. doi: 10.1111/jdv.15644. Epub 2019 May 10. No abstract available. PMID 31033034